CLINICAL TRIAL: NCT06935227
Title: Postoperative Outcomes of Steri-Strip Surgical Tape Use in Unilateral Ectropion Surgery: A Parallel-Controlled Clinical Trial
Brief Title: Steri-Strip Tape Use in Unilateral Ectropion Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Claudia Aristizábal (Other)
Responsible Party: Sponsor-Investigator, Claudia Aristizábal, Director, Sanitas University
Organization: Sanitas University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Steri-Strip Post-Surgery
Record Dates: First submitted 2025-04-11; First posted 2025-04-20 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Ectropion
MeSH Terms: conditions — Ectropion | interventions — Postoperative Period; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use Steri-Strip in post-surgery + standard care (Active Comparator): Within the first hour after unilateral ectropion surgery, Steri-Strip tapes (6 mm wide × 100 mm long, pack of 10 strips) will be applied to the operated eye. Six of these strips will be placed obliquely, hammock-style, 3 mm below the inferior orbital rim to direct the tension forces upward, using the lateral canthus of the operated eye as support. An additional strip will be placed horizontally, 2 mm above the orbital rim. The Steri-Strip tapes will be removed 8 days after surgery.
  Interventions: Other: Use Steri-Strip in post-surgery + standard care
- Standard care (Other): Standard care for ectropion surgery refers to the usual postoperative management provided without the use of additional supportive devices such as Steri-Strip tapes. It typically includes the application of ophthalmic antibiotic ointment, cold compresses, and instructions for eyelid hygiene.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Use Steri-Strip in post-surgery + standard care — Steri-strip will be maintained for 8 days postoperatively.
  Arms: Use Steri-Strip in post-surgery + standard care
Other: Standard care — Postoperative care recommendations.
  Arms: Standard care

SUMMARY:
Currently, the incidence of involutional and chronic eyelid disorders, such as ectropion, has been increasing, as human life expectancy has risen worldwide (more than 600 million people are aged ≥ 60 years). Ectropion is a common eyelid malposition that causes visual morbidity. It is characterized by eversion of the eyelid margin and has multiple etiologies.

Steri-Strip tapes have been used in some ophthalmologic procedures, such as blepharoplasties, where they help prevent infections by acting as a barrier method, are resistant enough to reduce the risk of wound dehiscence, simplify postoperative care, and allow for proper eyelid fissure closure. Their use has been recommended in patients with facial paralysis to prevent keratitis or exposure ulcers. However, current evidence is limited, as their use has only been documented in case series and letters to the editor. Therefore, a randomized controlled clinical trial is proposed to evaluate the postoperative outcomes of Steri-Strip tape use in unilateral ectropion surgery compared to standard postoperative management.

DETAILED DESCRIPTION:
This study will compare the use of Steri-Strip tape in unilateral ectropion surgery with standard postoperative care to assess cosmetic and functional outcomes in the adult population. Participants will be followed up at 8 and 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older who are scheduled to undergo unilateral ectropion surgery.

Exclusion Criteria:

* Underlying conditions associated with skin hyperlaxity, such as cutis laxa and Ehlers-Danlos syndrome.
* Skin diseases that predispose to cicatricial ectropion, such as ichthyosis, scleroderma, and psoriasis.
* Paralytic ectropion.
* Current use of oral isotretinoin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Eyelid position | Measurements will be taken in the immediate postoperative period (within the first hour) and at 30 days following surgery.
  This outcome will be assessed using the margin reflex distance 2 (MRD2), which will be measured in millimeters (mm) from the central corneal light reflex (Hirschberg reflex) to the center of the lower eyelid margin. If this measurement exceeds 5 mm, it suggests that the tapes did not provide adequate support.

SECONDARY OUTCOMES:
Surgical wound closure | This will be assessed on postoperative day 8
  This outcome will be evaluated using a slit lamp and defined as complete approximation of the wound edges. It will be recorded as a binary variable: Yes/No.
Visual axis obstruction secondary to peripalpebral edema | It will be assessed on postoperative day 8.
  This outcome will be evaluated using direct flashlight illumination. If a corneal light reflex is observed, it will indicate a clear visual axis.
Ocular surface symptoms | This outcome will be assessed on postoperative days 8 and 30.
  These symptoms are defined as the presence of ocular dryness, foreign body sensation, burning, or tearing. Each symptom will be recorded as present or absent. The presence of one or more of these symptoms will be interpreted as the occurrence of ocular surface symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Gomez, MD, Principal Investigator — Unisanitas
Locations (1):
- Oftalmosanitas, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No